CLINICAL TRIAL: NCT01282996
Title: Intraoperative Lung Protective Ventilation in Abdominal Surgery: A Randomized Controlled Study
Brief Title: Intraoperative Protective Ventilation in Abdominal Surgery (IMPROVE Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0087
Record Dates: First submitted 2011-01-18; First posted 2011-01-25 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Protective Lung Ventilation Using:; Low Tidal Volume (6-8 mL/kg Predicted Body Weight); PEEP of 6-8 cmH2O; Intraoperative RMs
Keywords: Mechanical ventilation; Postoperative pulmonary complications; Positive end-expiratory pressure; Protective lung ventilation; Alveolar recruitment maneuver; General anesthesia; Abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Other: Abdominal surgery — to compare the influence of a lung protective ventilation with conventional ventilation on postoperative complications following major abdominal surgery

SUMMARY:
The purpose of this study is to compare the influence of a lung protective ventilation with conventional ventilation on postoperative complications following major abdominal surgery.

DETAILED DESCRIPTION:
Postoperative complications are associated with a significant and quantifiable rate of both morbidity and mortality, increased length of hospital stay and cost of care. Intra-abdominal surgery, especially upper abdominal surgery, is an important risk factor of both pulmonary and extra-pulmonary complications. Up to 15-20% of patients will develop postoperative respiratory failure which may require respiratory support.

Recent data from both experimental and clinical studies suggested that, compared with conventional ventilation using high tidal volume (TV) without positive end-expiratory pressure (PEEP), intraoperative lung protective ventilation using low tidal volume, PEEP and recruitment maneuvers (RM) could reduce postoperative complications. Conventional ventilation promotes sustained cytokine production and could therefore contribute to development of lung injury with in patients with normal lungs. Conversely, lung protective ventilation was found to reduce pulmonary and systemic inflammation.

The primary objective is to compare a lung protective ventilation with conventional ventilation (high tidal volumes without PEEP) during abdominal surgery: 1- Conventional ventilation with TV of 10-12 mL/kg predicted body weight (PBW) without PEEP; 2- Protective lung ventilation with TV of 6-8 mL/kg PBW, PEEP of 6-8 cmH2O and RM.

Our hypothesis is that lung protective ventilation could reduce postoperative pulmonary and extra-pulmonary complications compared with conventional ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Planned intrabdominal surgery
* Expected duration ≥ 2 hours
* Age ≥ 40 yr (and <90 yr)
* Risk of postoperative pulmonary complications (Arozullah score ≥2)

Exclusion Criteria:

* Noninvasive ventilation in the last 30 days
* Recent history of pneumonia, ALI/ARDS (in the last 30 days)
* History of pulmonary resection
* History of neuromuscular disease
* Patient refusal

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint defined as incidence of major postoperative pulmonary (defined as pneumonia, need for noninvasive ventilation or need for invasive ventilation) and extrapulmonary (SIRS, sepsis and septic shock) complications | during the first seven days after surgery

SECONDARY OUTCOMES:
Major complications: postoperative hypoxemia, postoperative pneumonia, acute lung injury (ALI), acute respiratory distress syndrome (ARDS), pulmonary embolism | at day 15 after surgery
Minor complications : atelectasis, anastomotic leakage, intrabdominal abscess | at day 15 after surgery
Other postoperative complications (reintervention, wound abscess, ...) | at day 15 after surgery
Systemic level of marker of inflammation (C Reactive protein) | at day 15 after surgery
Postoperative complications at day 30 after surgery | at day 30 after surgery
Need for ICU admission | at day 30 after surgery
ICU length of stay | at day 30 after surgery
Hospital length of stay | at day 30 after surgery
Mortality | at day 30 after surgery
Plasma levels of the soluble form of the receptor for advanced glycation end-products (sRAGE), a marker of alveolar type I cell injury | before surgery, during the immediate postoperative period and on day 1, day 3 and day 7 after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Neuschwander A, Futier E, Jaber S, Pereira B, Eurin M, Marret E, Szymkewicz O, Beaussier M, Paugam-Burtz C. The effects of intraoperative lung protective ventilation with positive end-expiratory pressure on blood loss during hepatic resection surgery: A secondary analysis of data from a published randomised control trial (IMPROVE). Eur J Anaesthesiol. 2016 Apr;33(4):292-8. doi: 10.1097/EJA.0000000000000390. PMID 26716865
- [Derived] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482